CLINICAL TRIAL: NCT01425359
Title: A Phase 4, Randomized, Double-Blind, Placebo-Controlled, Parallel Study of Ranolazine in Subjects With Chronic Stable Angina and Coronary Artery Disease With a History of Type 2 Diabetes Mellitus
Brief Title: Type 2 Diabetes Evaluation of Ranolazine in Subjects With Chronic Stable Angina
Acronym: TERISA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-259-0133
Record Dates: First submitted 2011-08-24; First posted 2011-08-30 (Estimated); Results first posted 2014-11-04 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Angina Pectoris; Coronary Artery Disease; Type 2 Diabetes Mellitus
Keywords: Chronic angina; Angina pectoris; Coronary artery disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Angina Pectoris; Coronary Artery Disease; Diabetes Mellitus, Type 2 | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Qualifying phase: Participants will enter a 2-week washout period if needing to discontinue antianginal drugs (except beta-blockers) followed by placebo to match ranolazine (1 tablet twice daily) during a 4-week run-in period. Participants with at least 85% adherence to documentation requirements (angina frequency and sublingual nitroglycerin use) over the last 21 days of the placebo run-in period will be randomized to the treatment period.
  Treatment Period: Placebo to match ranolazine (Day 1: 1 tablet in the evening; Days 2-7: 1 tablet twice daily; 2 tablets twice daily thereafter) for up to 8 weeks.
  Interventions: Drug: Ranolazine placebo
- Ranolazine (Experimental): Qualifying phase: Participants will enter a 2-week washout period if needing to discontinue antianginal drugs (except beta-blockers) followed by placebo to match ranolazine (1 tablet twice daily) during a 4-week run-in period. Participants with at least 85% adherence to documentation requirements (angina frequency and sublingual nitroglycerin use) over the last 21 days of the placebo run-in period will be randomized to the treatment period.
  Treatment period: Ranolazine tablets (Day 1: 1 × 500 tablet in the evening; Days 2-7: 1 × 500 mg twice daily; 2 × 500 mg twice daily thereafter) for up to 8 weeks.
  Interventions: Drug: Ranolazine; Drug: Ranolazine placebo

INTERVENTIONS:
Drug: Ranolazine
  Other Names: Ranexa®
  Arms: Ranolazine
Drug: Ranolazine placebo

SUMMARY:
This study will evaluate the effect of ranolazine compared to placebo on the average weekly angina frequency in subjects with chronic stable angina and coronary artery disease (CAD) who have a history of type 2 diabetes mellitus (T2DM), and whether ranolazine can reduce the frequency of angina (chest pain) attacks, compared to a placebo. Subjects will be asked to record their daily angina episodes in a diary at the end of each study day. Ranolazine is approved for the treatment of chronic angina, and is not approved for the treatment of T2DM.

DETAILED DESCRIPTION:
Participants who meet the eligibility criteria at screening will enter a 4-to 6-week Qualifying Period. The allowed concomitant antianginal medication(s) must be maintained at a stable dose throughout the study. Participants will document the number of angina episodes, number of sublingual nitroglycerin doses taken, and a dyspnea score (on a scale from 1 to 5) on a daily basis in a diary. Participants eligible to stay in the study after the Qualifying Period will enter the 8-week double-blind dosing phase. Participants will have study visits at the end of Weeks 2 and 8. Participants will continue to document the number of angina episodes and number of sublingual nitroglycerin doses taken as well as a dyspnea score on a daily basis by the end of each day in their diary. In addition, participants will be called during Week 2 and at the end of Week 5 to encourage compliance. A safety follow-up phone call will be made 14 days after the last study visit or early discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Males and females aged at least 18 years
* At least a 3-month history of chronic stable angina triggered by physical effort and relieved by rest and/or sublingual nitroglycerin
* CAD documented by one or more of the following:

  1. Angiographic evidence of ≥ 50% stenosis of one or more major coronary arteries
  2. History of myocardial infarction (MI) documented by positive myocardial muscle creatine kinase (CK-MB) enzymes, troponins, or electrocardiogram (ECG) changes
  3. Cardiac imaging study or exercise test diagnostic for CAD
* Treatment with up to 2 antianginal therapies at a stable dose for at least 2 weeks prior to the Qualifying Period.
* Documented history of T2DM
* Willing to maintain stable tobacco usage habits throughout the study
* Willing to maintain stable activity levels throughout the study
* Females of childbearing potential must agree to utilize highly effective contraception methods from Screening throughout the duration of study treatment and for 14 days following the last dose of study drug.

Exclusion Criteria:

* New York Heart Association (NYHA) Class III and IV
* Acute coronary syndrome in the prior 2 months or planned coronary revascularization during the study period
* Stroke or transient ischemic attack within 6 months prior to Screening
* QTc > 500 milliseconds
* Uncontrolled hypertension (seated systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg)
* Systolic blood pressure < 100 mmHg
* Clinically significant hepatic impairment
* Prior treatment with ranolazine, or known hypersensitivity or intolerance to ranolazine
* Females who are breastfeeding
* Positive serum pregnancy test
* Participation in another investigational drug or device study within 1 month prior to Screening
* Current treatment with trimetazidine, ivabradine, or nicorandil. Subjects will need to discontinue these medications 2 weeks prior to the Qualifying Period.
* Current treatment with potent inhibitors of cytochrome (CYP)3A (eg, ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir, and saquinavir)
* Current treatment with CYP3A and P glycoprotein (Pgp) inducers (eg, rifampicin/rifampin, carbamazepine, and St. John's wort [Hypericum perforatum])
* Current treatment with CYP3A4 substrates with a narrow therapeutic range (eg, cyclosporine, tacrolimus, and sirolimus)
* Subjects taking simvastatin who cannot reduce the dose to 20 mg once daily or who cannot switch to another statin
* Current treatment with Class I or III antiarrhythmic medications
* History of illicit drug use or alcohol abuse within 1 year of Screening
* Any other conditions that, in the opinion of the investigator, are likely to prevent compliance with the study protocol or pose a safety concern if the subject participates in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 949 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yue, MD, Study Director — Gilead Sciences
Locations (132):
- United States (20):
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - Merced Heart Associates, Merced, California
  - Spectrum Clinical Research Institute, Inc, Moreno Valley, California
  - Sacramento Heart and Vascular Research Center, Sacramento, California
  - South Florida Research Solutions, LLC, Hollywood, Florida
  - Baptist Heart Specialist, Jacksonville, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Masters of Clinical Research, Inc., Augusta, Georgia
  - Columbus Cardiology Associates, Columbus, Georgia
  - Central Cardiology Associates, Elizabethtown, Kentucky
  - Research Integrity, LLC, Owensboro, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Clinical Trials Management, LLC, Mandeville, Louisiana
  - Endeavor Medical Research, PLC, Alpena, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Cross Country Cardiology, Edgewater, New Jersey
  - Kore CV Research, Jackson, Tennessee
  - Wellmont Cardiovascular Associates Heart Institute, Johnson City, Tennessee
  - Med-Tech Research, Houston, Texas
  - Humble Cardiology Associates, Humble, Texas
- Belarus (2):
  - State Institution "Gomel regional clinical hospital", Homyel
  - State Inst Rep Scientific and Practical center, Minsk
- Bulgaria (6):
  - Diagnostic Consultative Center, Ascendent Cardiological Out-Patient Office, Sofia
  - MHAT "Tsar Boris III", Sofia
  - National Cardiology Center, Cardiology Clinic - III, Sofia
  - MHAT "Vita", Cardiology Department, Sofia
  - UMHAT "Tsaritsa Yoanna" - ISUL, Cardiology Clinic, Sofia
  - Military Medical Academy, Clinic of Cardiology and Intesive Care, Sofia
- Canada (8):
  - Dr. Roger Labonté Professional Medicine Corp., Greater Sudbury, Ontario
  - SKDS Research Inc, Newmarket, Ontario
  - Aniol Gupta MD, Toronto, Ontario
  - Montréal General Hospital, Montreal, Quebec
  - High Desert Medical Group, Lancaster
  - Montreal Heart Institute, Montreal
  - London Road Diagnostic Clinic and Medical Centre, Ontario
  - Topsail Road Medical Clinic, St. John's
- Czechia (7):
  - Vojenska Nemocnice Brno, Brno
  - Cardiocentrum Kladno s.r.o., Kladno
  - Poliklinika Modrany - Kardiologie, Prague
  - Fakultní Nemocnice v Motole, Prague
  - Corintez s.r.o., Prague
  - Centrum klinického výzkumu, s.r.o., Príbram
  - Nemocnice Slaný, Slaný
- Georgia (7):
  - Tbilisi State Medical University Alexandre Aladashvili University Clinic, Tbilisi
  - Amtel Hospital First Clinical LLC, Tbilisi
  - Clinic "Guli", Tbilisi
  - Cardio-Reanimation Clinic LTD, Tbilisi
  - Emergency Cardiology Center by Academician G. Chapidze LTD, Tbilisi
  - Tbilisi Heart and Vascular Clinic LTD, Tbilisi
  - Multiprofile Clinical Hospital of Tbilisi #2 LTD, Tbilisi
- Germany (7):
  - Charité Campus Virchow Klinikum, Berlin
  - Städtische Kliniken Bielefeld, Bielefeld
  - Sankt Johannes-Hospital Dortmund, Dortmund
  - Universitätsklinikum Göttingen, Göttingen
  - Gemeinschaftspraxis fur Kardiologie, Heidelberg
  - Praxis Fur Innere Medizin Kardiologie, Pneumologic und Allergologie, Mannheim
  - Universitätsmedizin Mannheim, Mannheim
- Israel (6):
  - Barzilai Medical Center, Cardiology Dept., Ashkelon
  - Assaf Harofeh Medical Centre, Be’er Ya‘aqov
  - Shaare Zedek Medical Center, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
  - Tel Aviv Souraski Medical Center, Tel Aviv
- Poland (13):
  - Specjalistyczna Praktyka Lekarska Leszek Bryniarski, Krakow, Lesser Poland Voivodeship
  - NZOZ Revita Poradnia Kardiologiczna, Krakow, Lesser Poland Voivodeship
  - KO-MED Marek Konieczny, Puławy, Lublin Voivodeship
  - Instytut Kardiologii, Warsaw, Masovian Voivodeship
  - NZOZ Sródmiescie Sp z o.o., Gdynia, Pomeranian Voivodeship
  - Pomorskie Centra Kardiologiczne S.A., Gdansk
  - S.P. Specjalistyczny Szpital Zachodni im.JP II, Grodzisk Mazowiecki
  - Krakowski Szpital Specjalistyczny im.JPII, Krakow
  - Synexus SCM Sp. z o.o. Oddział w Warszawie, Warsaw
  - Centrum Badawcze Współczenej Terapii, Warsaw
  - Slaskie Centrum Chorób Serca w Zabrzu, Zabrze
  - MULTI-MED PLUS Sp. z o.o., Lódz, Łódź Voivodeship
  - Niepubliczny Zakład Opieki Zdrowotnej Przychodnia Zdrowia "Zadębie", Skierniewice, Łódź Voivodeship
- Russia (35):
  - City Hospital #38 named after Semashko N.A, Pushkin, Sankt-Peterburg
  - Altay Regional Cardiologycal Dispensary, Barnaul
  - "Chita State Medical Academy" Curative-Diagnostic Clinic department, Chita
  - Municipal Institution of Healthcare "Kemerovo Cardiology Dispensary", Kemerovo
  - Non-state Institution of healthcare "Department hospital on station Kemerovo of OAO "Russian Railway", Kemerovo
  - Medical centre "Delis", LLC, Kirovsk
  - Federal State Institution "National Research Center for Preventive Medicine", Moscow
  - State healthcare institution of Moscow "City Clinical hospital#15 named after O.M.Filatov", Moscow
  - State Healthcare institution of Moscow"Cardiology Dispensary #2", Moscow
  - First Moscow State Medical University I.M. Sechenov, Moscow
  - State Budget Educational Institution of High Professional Education First Moscow State Medical University... #1, Cardiology Clinic, Hospital Therapy Department, Moscow
  - Moscow City Clinical Hospital #51, Moscow
  - FGU Central Clinical Hospital with Polyclinic of President Administrative Department of RF, Moscow
  - Moscow State University of Medicine and Dentistry based on Moscow City Clinical Hospital #71, Moscow
  - City Clinical Hospital named after S.P.Botkin, Moscow
  - State Institution of Moscow Healthcare "City Clinical Hospital named after S.P. Botkin", Moscow
  - Moscow State Institution of Health "City Clinical Hospital #81", Moscow
  - Federal State Institution "Outpatient department #3" of President Management department of Russian Federation, Moscow
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Regional Clinical Hospital named after N.N.Burdenko, Penza
  - State Institution of Healthcare Perm Regional Hospital for War Veterans, Perm
  - State Healthcare Institution "Ryazan regional clinical cardiological dispensary", Ryazan
  - FGU Central Clinical Hospital with Polyclinic of President Administrative Department of RF, Saint Petersburg
  - Federal State Educational Institution of High Professional Education "Military Medical Academy n.a. S.M. Kirov" of the Ministry of Defence of Russia, Saint Petersburg
  - International Medical Center "SOGAZ", LLC, Saint Petersburg
  - State Healthcare institution "Municipal Out-patient Clinic #109", Saint Petersburg
  - Saint-Petersburg State Healthcare Institution, Saint Petersburg
  - Federal Heart, Blood and Endocrinology Centre n.a. Almazov, Saint Petersburg
  - Institution and Address: "Medical Research Institute", LLC, Saint Petersburg
  - State Institution of Healthcare "City Hospital #40 of Kurortniy administrative district, Saint Petersburg
  - "Clinical hospital named after S.R.Mirotvortsev", Saratov
  - Educational Institution of Higher Vocational Education "Smolensk State Medical Academy" on the base of Municipal Medicoprophylactic Institution "Hospital of Emergency Medical Care",, Smolensk
  - Autonomous healthcare institution of Voronezh region "Voronezh regional clinic consultative and diagnostic centre", Voronezh
  - Municipal Institution of Healthcare "Clinical Hospital #8 of Yaroslavl", Yaroslavl
  - Sverdlovsky Regional Clinical Hospital of Wars Veterans, Yekaterinburg
- Serbia (2):
  - Cardiology Clinic, Clinical Center Serbia, Belgrade
  - Institute of Cardiovascular Diseases, Kamenitz
- Slovakia (6):
  - ALIAN, s.r.o., Bardejov
  - Cardioconsult, s.r.o., Bratislava
  - Kardiovaskulárne centrum, s.r.o., Bratislava
  - CARDIO D&R, s.r.o., Košice
  - KARDIOMED, s.r.o., Lučenec
  - Kardiocentrum Nitra, s.r.o., Nitra
- Slovenia (3):
  - University Clinic of Respiratory and Allergic Diseases Golnik, Golnik
  - University Klinicni Center Ljubljana, Ljubljana
  - General Hospital Murska Sobota, Murska Sobota
- Ukraine (10):
  - Donetsk National Medical University, Department of Internal Medicine #1 based on Department of Emergency Cardiology and Rehabilitation of Institute of Urgent and Recovery Surgery named after V. K. Gusak, Donetsk
  - Central Clinical Hospital of Ukrzaliznitsia, Cardiology department, Kharkiv
  - Kharkiv Medical Academy of Postgraduate Education, Department of cardiology and functional diagnostics based on City Clinical Hospital #8, Department of Cardiology #2, Kharkiv
  - Central polyclinic of Pechersk district, Department of cardiology, Kyiv
  - Kyiv City Clinical Hospital #1, Department of Emergency Cardiology, Kyiv
  - Kyiv city clinical hospital #5, Kyiv
  - Department of Diabetology of National Medical Academy of Postgraduate Education named after P.L.Shupyk based on Day Time Hospital of Administration of Medical Service and Rehabilitation of "ARTEM" SHC, Kyiv
  - SI "Institute of Gerontology of AMS of Ukraine", Kyiv
  - Lviv National Medical University named after Danylo Halytsky, Department of Propaedeutics of Internal Medicine #1 based on Polyclinic Department of Municipal City Clinical Hospital #5, Lviv
  - SI Odessa Regional Cardiological Dispensary, Odesa

REFERENCES:
- [Derived] Arnold SV, Kosiborod M, Li Y, Jones PG, Yue P, Belardinelli L, Spertus JA. Comparison of the Seattle Angina Questionnaire With Daily Angina Diary in the TERISA Clinical Trial. Circ Cardiovasc Qual Outcomes. 2014 Nov;7(6):844-50. doi: 10.1161/CIRCOUTCOMES.113.000752. Epub 2014 Sep 23. PMID 25249560
- [Derived] Roubinian NH, Escobar GJ, Liu V, Gardner MN, Carson JL, Kleinman SH, Murphy EL; NHLBI Recipient Epidemiology and Donor Evaluation Study (REDS-III). Decreased red blood cell use and mortality in hospitalized patients. JAMA Intern Med. 2014 Aug;174(8):1405-7. doi: 10.1001/jamainternmed.2014.2889. No abstract available. PMID 24978650
- [Derived] Kosiborod M, Arnold SV, Spertus JA, McGuire DK, Li Y, Yue P, Ben-Yehuda O, Katz A, Jones PG, Olmsted A, Belardinelli L, Chaitman BR. Evaluation of ranolazine in patients with type 2 diabetes mellitus and chronic stable angina: results from the TERISA randomized clinical trial (Type 2 Diabetes Evaluation of Ranolazine in Subjects With Chronic Stable Angina). J Am Coll Cardiol. 2013 May 21;61(20):2038-45. doi: 10.1016/j.jacc.2013.02.011. Epub 2013 Mar 10. PMID 23500237

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 116 study sites in North America, Europe, and Asia. The first participant was screened on 05 October 2011. The last participant observation occurred on 25 October 2012.
Pre-assignment Details: 1142 participants entered the qualifying period.
Groups:
- Placebo: Qualifying phase: Participants entered a 2-week washout period if needed to discontinue antianginal drugs (except beta-blockers) followed by placebo to match ranolazine (1 tablet twice daily) during a 4-week run-in period. Participants with at least 85% adherence to documentation requirements (angina frequency and sublingual nitroglycerin use) over the last 21 days of the placebo run-in period were randomized to the treatment period.
  Treatment Period: Placebo to match ranolazine (Day 1: 1 tablet in the evening; Days 2-7: 1 tablet twice daily; 2 tablets twice daily thereafter) for up to 8 weeks.
- Ranolazine: Qualifying phase: Participants entered a 2-week washout period if needed to discontinue antianginal drugs (except beta-blockers) followed by placebo to match ranolazine (1 tablet twice daily) during a 4-week run-in period. Participants with at least 85% adherence to documentation requirements (angina frequency and sublingual nitroglycerin use) over the last 21 days of the placebo run-in period were randomized to the treatment period.
  Treatment period: Ranolazine tablets (Day 1: 1 × 500 tablet in the evening; Days 2-7: 1 × 500 mg twice daily; 2 × 500 mg twice daily thereafter) for up to 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Ranolazine
Started | 476 | 473
Completed | 457 | 451
Not Completed | 19 | 22
Not completed — Randomized but Not Treated | 2 | 3
Not completed — Adverse Event | 9 | 8
Not completed — Revascularization | 0 | 1
Not completed — Death | 0 | 1
Not completed — Unsatisfactory Response | 1 | 0
Not completed — Protocol Violation | 1 | 2
Not completed — Subject Withdrew Consent | 1 | 2
Not completed — Investigator's Discretion | 2 | 0
Not completed — Did Not Meet Qualifying Criteria | 3 | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: randomized participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ranolazine | Total
Number analyzed (Participants) | 474 | 470 | 944
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8.5) | 63 (8.6) | 64 (8.5)
Age, Customized [Number; unit: participants]
  < 65 years | 249 | 264 | 513
  65 - 74 years | 170 | 160 | 330
  ≥ 75 years | 55 | 46 | 101
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 180 | 362
  Male | 292 | 290 | 582
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1 | 1 | 2
  Black or African American | 2 | 5 | 7
  White | 471 | 464 | 935
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 464 | 462 | 926
  Not Reported | 3 | 3 | 6
  Unknown | 2 | 1 | 3
Region of Enrollment [Number; unit: participants] — All randomized participants were analyzed for region of enrollment (placebo, n = 476; ranolazine, n = 473).
  participants
    United States | 12 | 15 | 27
    Belarus | 1 | 0 | 1
    Serbia | 3 | 2 | 5
    Slovenia | 0 | 1 | 1
    Slovakia | 12 | 9 | 21
    Ukraine | 53 | 69 | 122
    Israel | 10 | 14 | 24
    Russian Federation | 281 | 263 | 544
    Czech Republic | 3 | 6 | 9
    Canada | 2 | 1 | 3
    Poland | 53 | 40 | 93
    Bulgaria | 9 | 11 | 20
    Georgia | 36 | 40 | 76
    Germany | 1 | 2 | 3
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.1 (4.90) | 31.3 (5.01) | 31.2 (4.96)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent HbA1c in blood] | 7.3 (1.53) | 7.3 (1.50) | 7.3 (1.52)

OUTCOME MEASURES:

1. Primary Outcome: Average Weekly Angina Frequency Over the Last 6 Weeks of Treatment
Description: Average weekly angina frequency was defined as the total number of angina episodes reported during the last 6 weeks of treatment divided by 6 weeks.
  For subjects who terminated with less than 6 weeks of treatment, frequency was calculated as the total number of angina episodes reported during the treatment period divided by the subject's actual duration of treatment.
Time Frame: 6 weeks
Population: Full Analysis Set (FAS): randomized participants who received at least 1 dose of randomized study drug with at least 1 postbaseline primary efficacy measurement and did not have any major eligibility violations. Participants were included in the FAS if they did not discontinue study drug prior to Day 14.
Measure: Mean (Standard Deviation); unit: angina attacks per week
Arm/Group | Placebo | Ranolazine
Number analyzed (Participants) | 465 | 462
angina attacks per week | 5.2 (4.73) | 4.5 (4.32)
Statistical Analysis 1: Comparison: Placebo vs Ranolazine; Test type: Superiority or Other; p = 0.008, Generalized linear model — Angina frequency was compared by fitting a generalized linear model with log link and negative binomial distribution response

2. Secondary Outcome: Average Weekly Frequency of Sublingual Nitroglycerin Use Over the Last 6 Weeks of Treatment
Description: Average weekly frequency of sublingual nitroglycerin use was defined as the total number reported during the last 6 weeks of treatment divided by the duration corresponding to the last 6 weeks of treatment.
Time Frame: 6 weeks
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: nitroglycerin uses per week
Arm/Group | Placebo | Ranolazine
Number analyzed (Participants) | 465 | 462
nitroglycerin uses per week | 3.6 (5.35) | 2.9 (4.34)
Statistical Analysis 1: Comparison: Placebo vs Ranolazine; Test type: Superiority or Other; p = 0.003, Generalized linear model — Sublingual nitroglycerin use frequency was compared by fitting a generalized linear model with log link and negative binomial distribution response

3. Secondary Outcome: Percentage of Weeks Participants Achieved at Least a 50% Reduction in Angina Frequency
Description: For each participant, the percentage of the last 6 weeks on treatment during which the angina frequency was less than or equal to 50% of the baseline average weekly angina frequency was determined.
Time Frame: 6 weeks
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of weeks
Arm/Group | Placebo | Ranolazine
Number analyzed (Participants) | 462 | 460
percentage of weeks | 41 (36) | 46 (35)

4. Secondary Outcome: Percentage of the Last 6 Weeks on Treatment During Which the Angina Frequency Was ≤ 50% of the Baseline Average Weekly Angina Frequency
Time Frame: 6 weeks
Population: Full Analysis Set
Measure: Mean (Standard Error); unit: percentage of weeks
Arm/Group | Placebo | Ranolazine
Number analyzed (Participants) | 465 | 462
percentage of weeks | 50 (1.4) | 54 (1.3)

5. Secondary Outcome: Change From Baseline in the Short-Form 36® (SF-36) Mental and Physical Component Scores
Description: The range of each health domain score is 0-100, with 0 indicating a poorer health state and 100 indicating a better health state. An increase in score indicates an improvement in health state. Participants were asked to complete the survey at randomization (prior to receiving treatment), and at end of treatment visit (Week 8) or early study drug discontinuation or early termination visit. The survey asked participants for responses specific to the preceding 4 weeks prior to completing the survey.
Time Frame: Up to 8 weeks
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Qualifying Phase: Participants Entered a 2-week Washout Period: Qualifying phase: Participants entered a 2-week washout period if needed to discontinue antianginal drugs (except beta-blockers) followed by placebo to match ranolazine (1 tablet twice daily) during a 4-week run-in period. Participants with at least 85% adherence to documentation requirements (angina frequency and sublingual nitroglycerin use) over the last 21 days of the placebo run-in period were randomized to the treatment period.
  Treatment period: Ranolazine tablets (Day 1: 1 × 500 tablet in the evening; Days 2-7: 1 × 500 mg twice daily; 2 × 500 mg twice daily thereafter) for up to 8 weeks.
Arm/Group | Placebo | Qualifying Phase: Participants Entered a 2-week Washout Period
Number analyzed (Participants) | 460 | 456
units on a scale
  Mental Component Score | 1.2 (0.37) | 1.0 (0.39)
  Physical Component Score | 1.9 (0.25) | 2.8 (0.26)

6. Secondary Outcome: Patient's Global Impression of Change (PGIC) Scale Score
Description: The PGIC was completed at the end of treatment/last visit.The PGIC scale measures the change in the participant's overall status since the beginning of the study on a scale ranging from 1 (no change or worse) to 7 (very much improved).
Time Frame: 8 weeks
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ranolazine
Number analyzed (Participants) | 461 | 457
units on a scale | 3.9 (0.07) | 4.0 (0.07)

ADVERSE EVENTS:
Time Frame: Baseline to Day 56 plus 30 days
Description: Safety Analysis Set: randomized participants who received at least one dose of study treatment.
Arm/Group | Placebo | Ranolazine
Serious Adverse Events (participants affected / at risk) | 20/474 | 16/470
Other Adverse Events (participants affected / at risk) | 0/474 | 0/470
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=474) | Ranolazine (N=470)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 2
Angina unstable (Cardiac disorders) | 1 | 3
Angina pectoris (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Chest pain (General disorders) | 1 | 2
Sudden cardiac death (General disorders) | 0 | 1
Thrombosis in device (General disorders) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 1
Cervical myelopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years